CLINICAL TRIAL: NCT04797052
Title: Prefrontal EEG Early Detection of Delirium in Older Adults
Brief Title: EEG Detection of Delirium
Acronym: VEEGilance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: TransMedTech Institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20.377
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Post Operative Delirium
Keywords: Post operative delirium; Older Adults; Electroencephalography
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Intervention Model Description: Prospective observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post operative patients (Experimental): Post operative patient in orthopedic and digestive surgery
  Interventions: Device: Prefrontal EEG (VEEGix by NeuroServo)

INTERVENTIONS:
Device: Prefrontal EEG (VEEGix by NeuroServo) — Prefrontal EEG reading

SUMMARY:
VEEGix is a portable device developed by NeuroServo for simplifying electroencephalograms at the bedside. It is an easy-to-use device that only requires the operator to place an adhesive strip of electrodes on the patient's forehead, connected to the device. The goal of this study is to determine EEG thresholds for the diagnostic of delirium.

Methods : This prospective observational study includes patients undergoing orthopedic or degestive surgery. Each subject will have an EEG reading before surgery and twice daily after surgery until discharge or up to 5 days. Patients will be monitored for post operative delirium using the 3D-Confusion Assessment Method. Delirium diagnostic will be confirmed by a geriatrician. EEG relative power reading will be compared between patient with and without a delirium diagnostic.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older
* Had a orthopedic or digestive surgery
* Good undersanding of French or English
* Consent to participate in the study

Exclusion Criteria:

* History of seizure or epilepsia
* Structural brain damage
* intelectual deiciency
* Severe major neurocognitive disorder
* incapacity to respond to the questionnaire
* Hospitalised in intensive care or intubated

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 234 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Difference of relative power of delta and theta brain waves | up to five days after the operation
  Difference between group with and without delirium

SECONDARY OUTCOMES:
Difference of relative power of beta and alpha brain waves | up to five days after the operation
  Difference between group with and without delirium
describe the presence of artefacts | up to five days after the operation
  Examine the EEG reading for artefacts

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada